CLINICAL TRIAL: NCT00554541
Title: Lower Extremity Venous Hemodynamics in Obese Patients Without Clinically Significant Venous Disease
Status: Terminated | Type: Observational
Why Stopped: Lack of study subjects
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Heather Gornik, Principal Investigator, The Cleveland Clinic
Other Study IDs: 07-617
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Obesity; Peripheral Arterial Disease
MeSH Terms: conditions — Obesity; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal Body-Mass: BMI Index: 18.5-24.9 Ankle Brachial Index Venous physiologic study
  Interventions: Other: Ankle Brachial Index Venous physiologic study
- Obese Body-Mass: BMI Index: 30.0-39.9 Ankle Brachial Index Venous physiologic study
  Interventions: Other: Ankle Brachial Index Venous physiologic study
- Morbidly Obese Body-Mass: BMI Index: ≥ 40 Ankle Brachial Index Venous physiologic study
  Interventions: Other: Ankle Brachial Index Venous physiologic study

INTERVENTIONS:
Other: Ankle Brachial Index Venous physiologic study — Assessment of lower extremity venous disease
  Other Names: ABI

SUMMARY:
This research project is investigating the relationship between body weight and function of the leg veins using a special non-invasive technique known as venous plethysmography.

DETAILED DESCRIPTION:
Disease of the veins include blood clots, varicose veins, leg swelling, and sores on the legs. Venous disease is more common in overweight patients, but little is known as to why this is the case. This research project is investigating the relationship between body weight and function of the leg veins using a special non-invasive technique known as venous plethysmography. We hope to investigate the reason for the relationship between body weight and higher risk of vein problems.

Approximately 45 people will take part in this study. Patients will be recruited from among three groups: normal weight people, overweight people, and obese people.

Resting ankle-brachial index will be measured in both lower extremities to exclude the presence of peripheral arterial disease. Venous physiologic study using air plethysmography with positional maneuvers will be performed. Parameters to be measured will be outflow time, passive draining and refill time, and exercise venous plethysmography. All studies will be performed with the Phlebotest system (Osborn Medical).

All study procedures will be done during one visit, and no further follow-up is required.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-60 years old
* BMI within one of three strata (Normal: 18.5-24.9, Obese: 30.0-39.9, Morbidly Obese: ≥ 40)

Exclusion Criteria:

* Prior diagnosis of chronic venous insufficiency or venous stasis ulceration
* Prior diagnosis of lymphedema
* Significant lower extremity edema as determined by study investigators. Lipidemia (in the absence of venous or lymphatic related edema) is acceptable.
* Varicose veins (subcutaneous dilated vein > 3 mm in diameter measured in upright position). Subjects with telangiectasias and/or mild reticular veins will be eligible (CEAP C1)
* Patients who have been prescribed compression stockings by a health care provider at any time in the past, aside from prophylactic use during prior hospitalization to prevent VTE
* Patients who have undergone any procedure for treatment of lower extremity varicose veins, including: sclerotherapy, venous ablation, phlebectomy, or a stripping procedure
* History of DVT or SVT
* Pregnancy
* Active malignancy
* Documented hypercoagulable state
* Body weight exceeds weight limit of the venous air plethysmograph chair equipment (approximately 375 lbs)
* Clinical diagnosis of lower extremity peripheral arterial disease or abnormal ankle-brachial index (ABI) in either lower extremity
* History of surgical intervention involving pelvis or lower extremities
* Pelvic or lower extremity radiation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients of the Cleveland Clinic Foundation.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is to investigate the reason for the relationship between body weight and higher risk of venous problems. | single time point

CONTACTS AND LOCATIONS:
Overall Officials: Heather Gornik, MD, RVT, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No